CLINICAL TRIAL: NCT02953938
Title: A 12-month, Phase IV, Open-label, Randomized, Active Controlled, 2-arm, Multicenter Study Assessing the Efficacy and Safety of Intravitreal Ranibizumab Combined With Grid&Direct Short Pulse Laser Photocoagulation Versus a PRN Ranibizumab Monotherapy in Japanese Patients With Macular Edema Secondary to Branch Retinal Vein Occlusion (BRVO)
Brief Title: Study to Show a Superior Benefit in Terms of Reduction of Ranibizumab Injections in Patients Receiving Ranibizumab Plus Laser Photocoagulation Combination Therapy Without Loss of Efficacy and Safety
Acronym: ZIPANGU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002EJP09
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Macular Edema Secondary to Branch Retinal Vein Occlusion (BRVO)
Keywords: Ranibizumab; Grid&Direct short pulse laser photocoagulation; Macular edema; Branch retinal vein occlusion; BRVO; BCVA; CSFT; pro re nata
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Ranibizumab

STUDY DESIGN:
Intervention Model Description: Phase IV, randomized, open-label, active-controlled, 2-arm, multicenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mono therapy (Active Comparator): ranibizumab alone
  Interventions: Biological: Ranibizumab
- combination therapy (Experimental): ranibizumab with Grid&Direct short pulse laser photocoagulation
  Interventions: Biological: Ranibizumab; Radiation: Grid&Direct short pulse laser photocoagulation

INTERVENTIONS:
Biological: Ranibizumab — Ranibizumab is a biologic and known anti-VEGF (vascular endothelial growth factor) medication approved for treatment of ME (Macular Edema) due to RVO (Retinal Vein occlusion)
  0.5 mg ranibizumab applied one + PRN as intravitreal injection of 0.05 mL, with or without laser treatment
  Other Names: RFB002E
Radiation: Grid&Direct short pulse laser photocoagulation — Grid&Direct short pulse laser photocoagulation is a kind of laser treatment to retina within vascular arcades and used to suppress macular edema
  Arms: combination therapy

SUMMARY:
This is a Phase IV, randomized, open-label, active-controlled, 2-arm, multicenter study. The primary objective was assessed by the difference in the mean number of ranibizumab injections applied up to Month 11 between the 2 treatment arms. Patients were randomized in a 1:1 ratio to 1 of the 2 treatment arms; i.e. Arm 1 ranibizumab monotherapy, Arm 2 ranibizumab with Grid&Direct short pulse laser photocoagulation combination therapy. There were 3 periods in this study: Screening Period (visit 1), Treatment Period (visit 2 to Visit 13) and Follow-up Period (visit 14). In addition to screening and Baseline (visit 2), there were monthly visits from Month 1 to Month 12. This study included male and female patients (≥20 years old) diagnosed with visual impairment due to ME secondary to BRVO.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of visual impairment exclusively due to ME secondary to BRVO
* Best-corrected visual acuity score at Screening and Baseline (Day 1) between 0.5 and 0.05 decimal (i.e., between 73 and 19 letters in Early Treatment Diabetic Retinopathy Study (ETDRS) testing) with Landolt C charts inclusively (i.e., approximate logarithm of the minimum angle of resolution (logMAR) units of 0.3 to 1.30).
* At Baseline (Day1), a maximum BCVA gain of 0.2 units logMAR conversion inclusively from screening is allowed as long as the BCVA score does not exceed the upper limit of 0.3 units logMAR.
* Increased central subfoveal thickness (> 300 µm at Baseline (Day 1) when measured by SD-OCT)
* Duration of vision deterioration ≤6 months (determined by self-report) at screening

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Stroke or myocardial infarction less than 3 months before Screening
* Uncontrolled blood pressure defined as systolic value of >160 mm Hg or diastolic value of >100 mm Hg at Screening or Baseline (Day 1) Antihypertensive treatment can be initiated and must be taken for at least 30 days after which the patient can be assessed for study eligibility a second time
* Any active periocular or ocular infection or inflammation (e.g., blepharitis, conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) at the time of Screening or Baseline (Day 1) in either eye
* Uncontrolled glaucoma (intraocular pressure (IOP) ≥30 mm Hg on medication or according to investigator's judgment) at the time of Screening or Baseline (Day 1) or diagnosed within 6 months before Baseline (Day 1) in either eye
* Neovascularization of the iris or neovascular glaucoma in the study eye
* Use of any systemic anti-VEGF drugs within 6 months before Baseline (Day1) (e.g., sorafenib (Nexavar®), sunitinib (Sutent®), bevacizumab (Avastin®), ziv-aflibercept (ZALTRAP®))
* Treatment (or anticipated treatment in the fellow eye for non-RVO indications during the study) with any anti-angiogenic drugs (including any anti-VEGF agents) within 3 months before Baseline (Day1) in fellow eye or before Baseline (Day 1) in the study eye (e.g., pegaptanib (Macugen®), ranibizumab (Lucentis®), bevacizumab (Avastin®), and aflibercept (EYLEA®))
* Panretinal laser photocoagulation within 1 month before Baseline (Day1) or anticipated or scheduled within the next 12 months (Study periods) following Baseline (Day1) in the study eye
* Any giving of focal or grid laser photocoagulation before Baseline (Day1) in the study eye
* Use of intra- or periocular corticosteroids (including sub-Tenon) within 3 months before Screening in the study eye.
* Any use of intraocular corticosteroid implants (e.g., dexamethasone (Ozurdex®), fluocinolone acetonide (Iluvien®)) in the study eye

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Japan (7):
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Tsu, Mie-ken
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Mitaka, Tokyo
  - Novartis Investigative Site, Hokkaido

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 73 patients were screened and 59 were randomized on a 1:1 ratio to the ranibizumab group (29 patients) and ranibizumab with laser group (30 patients). Of the randomized patients, 56 (94.9%) completed the study and 11 months of treatment. 3 (5.1%) discontinued both study and study treatment: 2 (3.4%) withdrew consent and 1 (1.7%) had adverse event
Pre-assignment Details: Below is the participant flow of Randomized patients
Groups:
- Ranibizumab 0.5 mg: 0.5 mg ranibizumab applied one + PRN as intravitreal injection of 0.05 mL
- Ranibizumab 0.5 mg and Laser: 0.5 mg ranibizumab applied one + PRN as intravitreal injection of 0.05 mL with the laser treatment
Period: Overall Study
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg and Laser
Started | 29 | 30
Completed (Completed Study Prior to 12 Months) | 28 | 28
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg and Laser | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.91) | 66.7 (9.83) | 66.8 (9.78)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 12 | 11 | 23
  >=65 years | 17 | 19 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 19 | 29
  Male | 19 | 11 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mean Number of Ranibizumab Injections
Description: Number of ranibizumab treatments from Day 1 to Month 11 using full analysis set (observed) based on a stratified Cochran-Mantel-Haenszel (CMH) test. Stratification was done based on categories of baseline decimal VA (<0.3, or =>0.3). Difference of mean number of injections, 95% confidence interval (CI) of difference and one-sided p-value of the CMH test was reported. Analysis was conducted within the FAS with observed data.
  Stratification was based on baseline visual acuity on logMAR scale (<0.52, >=0.52). Test was one-sided.
Time Frame: Month 1 through Month 12
Population: Randomized Set, i.e.; all randomized patients.
Measure: Mean (Standard Deviation); unit: number of injections
Groups:
- Ranibizumab 0.5 mg Laser: 0.5 mg ranibizumab applied one + PRN as intravitreal injection of 0.05 mL with the laser treatment.
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg Laser
Number analyzed (Participants) | 29 | 30
number of injections | 4.3 (2.51) | 4.1 (2.41)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Ranibizumab 0.5 mg Laser; Test type: Superiority; p = 0.3680, Cochran-Mantel-Haenszel; Mean Difference (Net) = -0.21, 95% CI 2-sided [-1.49 to 1.07], Standard Deviation 0.64

2. Secondary Outcome: The Mean Change in Best Corrected Visual Acuity (BCVA) Using Decimal Chart and Early Treatment Diabetic Retinopathy Study (ETDRS) Compared to Baseline
Description: Summary of BCVA (letters) absolute value and change from Baseline at Month 12 in the study eye - full analysis set (LOCF) was based on an analysis of variance (ANOVA) model with treatment group, and stratification factors. Stratification was done based on categories of baseline decimal VA (<0.3, or =>0.3). The analyses was conducted within the FAS using the LOCF approach
  Stratification was based on baseline visual acuity on logMAR scale (<0.52, >=0.52). Test was one-sided.
Time Frame: Month 1 through Month 12 (for ETDRS: Month 6 and Month 12)
Population: The Full Analysis Set (FAS) consisted of all randomized patients who received at least one administration of ranibizumab injection.
Measure: Mean (Standard Deviation); unit: letters read correctly
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg Laser
Number analyzed (Participants) | 29 | 30
letters read correctly
  baseline | 52.86 (13.384) | 54.03 (9.828)
  month 12 | 74.83 (9.740) | 69.59 (8.842)
  change from baseline to month 12 | 21.97 (14.749) | 15.00 (10.296)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Ranibizumab 0.5 mg Laser; Test type: Superiority; p = 0.0349, ANOVA; Mean Difference (Final Values) = -6.58, 95% CI 2-sided [-12.67 to -0.48], Standard Deviation 3.042

3. Secondary Outcome: The Mean Change in BCVA From Month 1 Through Month 12 Compared to Baseline (Day 1) by the Treatment Arms
Description: Summary of BCVA (logMAR) absolute value and change from Baseline at Month 12 in the study eye - full analysis set (LOCF) was based on an analysis of variance (ANOVA) model with treatment group, and stratification factors. Stratification was based on baseline visual acuity (< 0.52, >= 0.52). The analyses was conducted within the FAS using the LOCF approach
Time Frame: Month 1 through Month 12
Population: FAS
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg Laser
Number analyzed (Participants) | 29 | 30
logMAR
  baseline | 0.553 (0.2276) | 0.558 (0.1719)
  month12 | 0.075 (0.1909) | 0.143 (0.1682)
  change from baseline to month 12 | -0.478 (0.2586) | -0.413 (0.1969)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Ranibizumab 0.5 mg Laser; Test type: Superiority; p = 0.2707, ANOVA; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.045 to 0.158], Standard Deviation 0.051

4. Secondary Outcome: BCVA (Letters) Number and Proportion of Patients With a BCVA Improvement vs. Baseline, Loss Less Than 15 Letters, or Attainment of Greater Than or Equal to 85 Letters at Month 6 and at Month 12 in the Study Eye
Description: Endpoints related to the number and proportion of patients with BCVA letter gain or loss from Baseline (Day1) was analyzed via stratified CMH test with stratification factors as described in primary model. The mean (SD) average (per patient) BCVA (logMAR) change from Baseline through Month 12
  Summary of BCVA (logMAR) mean average change from Baseline from Month 1 through Month 12 in the study eye
Time Frame: Month 6 and Month 12
Population: Full Analysis Set (FAS) consisted of all randomized patients who received at least one administration of ranibizumab injection
Measure: Count of Participants; unit: Participants
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg Laser
Number analyzed (Participants) | 29 | 30
Participants
  Month 6 - BCVA improvement of >=1: number analyzed (Participants) | 29 | 29
  Month 6 - BCVA improvement of >=1 | 27 | 24
  month 6 - BCVA improvement of >=5: number analyzed (Participants) | 29 | 29
  month 6 - BCVA improvement of >=5 | 26 | 21
  month 6 - BCVA improvement of >=10: number analyzed (Participants) | 29 | 29
  month 6 - BCVA improvement of >=10 | 22 | 16
  Month 6 - BCVA improvement of >=15: number analyzed (Participants) | 29 | 29
  Month 6 - BCVA improvement of >=15 | 17 | 12
  Month 6 - BCVA improvement of >=30: number analyzed (Participants) | 29 | 29
  Month 6 - BCVA improvement of >=30 | 4 | 1
  month 6 Score >=73: number analyzed (Participants) | 29 | 29
  month 6 Score >=73 | 12 | 10
  month 6 Score >=80: number analyzed (Participants) | 29 | 29
  month 6 Score >=80 | 8 | 2
  month 6 Score >=85: number analyzed (Participants) | 29 | 29
  month 6 Score >=85 | 3 | 1
  month 6 loss of <15: number analyzed (Participants) | 29 | 29
  month 6 loss of <15 | 28 | 29
  Month 12 - BCVA improvement of >=1: number analyzed (Participants) | 29 | 29
  Month 12 - BCVA improvement of >=1 | 27 | 28
  Month 12 - BCVA improvement of >=5: number analyzed (Participants) | 29 | 29
  Month 12 - BCVA improvement of >=5 | 27 | 25
  Month 12 - BCVA improvement of >=10: number analyzed (Participants) | 29 | 29
  Month 12 - BCVA improvement of >=10 | 24 | 18
  Month 12 - BCVA improvement of >=15: number analyzed (Participants) | 29 | 29
  Month 12 - BCVA improvement of >=15 | 21 | 15
  Month 12 - BCVA improvement of >=30: number analyzed (Participants) | 29 | 29
  Month 12 - BCVA improvement of >=30 | 9 | 3
  month 12 Score >=73: number analyzed (Participants) | 29 | 29
  month 12 Score >=73 | 20 | 10
  month 12 Score >=80: number analyzed (Participants) | 29 | 29
  month 12 Score >=80 | 8 | 13
  month 12 Score >=85: number analyzed (Participants) | 29 | 29
  month 12 Score >=85 | 4 | 0
  month 12 Loss of <15: number analyzed (Participants) | 29 | 29
  month 12 Loss of <15 | 29 | 29

5. Secondary Outcome: The Mean Change in Change in Central Subfield Foveal Thickness (CSFT) From Month 1 Through Month 12 Compared to Baseline (Day1) by the Treatment Arms
Description: The mean change in investigator-assessed CSFT from Month 1 through Month 12 was compared to Baseline (Day1) by the treatment arms. The analyses at each visit was based on an analysis of variance (ANOVA) model as analogous to BCVA. The analyses was conducted within the FAS using the Last-Observation-Carried-Forward (LOCF) approach
Time Frame: Month 1 through Month 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg Laser
Number analyzed (Participants) | 29 | 30
mm
  baseline | 563.3 (146.92) | 553.3 (182.39)
  month 12 | 257.0 (43.44) | 285.1 (82.80)
  change in baseline from month 12 | -306.3 (164.35) | -261.3 (180.23)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Ranibizumab 0.5 mg Laser; Test type: Superiority; p = 0.7602, ANOVA; Mean Difference (Final Values) = 11.32, 95% CI 2-sided [-62.65 to 85.28]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected for the maximum duration of treatment and follow up for a participant per protocol for approximately 12 months.
Description: All cause mortality (deaths) was collected from First Patient First Visit (FPFV) to Last Patient Last Visit (LPLV) up to a maximum of 12 months
Groups:
- Ranibizumab 0.5 mg+ Laser: 0.5 mg ranibizumab applied one + PRN as intravitreal injection of 0.05 mL with the laser treatment.
- Total: Total
Arm/Group | Ranibizumab 0.5 mg | Ranibizumab 0.5 mg+ Laser | Total
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30 | 0/59
Serious Adverse Events (participants affected / at risk) | 1/29 | 2/30 | 3/59
Other Adverse Events (participants affected / at risk) | 16/29 | 15/30 | 31/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=29) | Ranibizumab 0.5 mg+ Laser (N=30) | Total (N=59)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Putamen haemorrhage (Nervous system disorders) | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=29) | Ranibizumab 0.5 mg+ Laser (N=30) | Total (N=59)
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 1
Corneal erosion (Eye disorders) | 0 | 1 | 1
Dry eye (Eye disorders) | 1 | 1 | 2
Keratitis (Eye disorders) | 1 | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 1 | 1
Photopsia (Eye disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 3
Feeling abnormal (General disorders) | 0 | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 1 | 2
Influenza (Infections and infestations) | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 6 | 5 | 11
Periodontitis (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Intraocular pressure increased (Investigations) | 0 | 3 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 2
Dysarthria (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 3 | 0 | 3
Hemiplegia (Nervous system disorders) | 0 | 1 | 1
Migraine (Nervous system disorders) | 0 | 1 | 1
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypertension (Vascular disorders) | 2 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreement with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publications of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-01-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT02953938/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/38/NCT02953938/SAP_001.pdf